CLINICAL TRIAL: NCT03338452
Title: The Safety and Effects on Whole Organism of Low Energy Ketogenic Diet for Weight Loss in Obese Subjects
Brief Title: Low Energy Ketogenic Diet in Obese Subjects - the Impact on Whole Organism
Acronym: KETO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, Assist. prof. dr. sc., University of Primorska
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEKD2017
Record Dates: First submitted 2017-10-27; First posted 2017-11-09 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Obesity
Keywords: ketogenic diet; body composition; metabolism; body dissatisfaction; cognition
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Longitudinal intervention study with repeated measurements. Participants will be subjected to a 12-week low energy ketogenic diet (LEKD) and requested not to change their physical activity levels throughout the study.
  The participants will underwent a series of tests and consultations at baseline (prior to the start of the intervention), and after 1, 2, 4, 8 , and 12 weeks of LEKD intervention. At the end of each time points, body weight and composition will be measured in the fasting state, food and exercise diaries checked by a dietitian and a kinesiologist and discussed with the participants, psychological and cognitive tests will be performed by a psychologist. At the same time-points, different serum analyses will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- participants (Experimental): The participants will be subjected to low energy ketogenic diet.
  Interventions: Behavioral: Low energy ketogenic diet

INTERVENTIONS:
Behavioral: Low energy ketogenic diet — Low energy ketogenic diet lasting 12 weeks with a previous preparation period including detailed instructions during classes and individual counselling by a dietitian. Participants were provided with a list of suitable foods with very low carbohydrate content. Furthermore, the subjects shared cooking recipes and links to helpful webpages. They were free to follow a KD according to their personal preferences but limit their carbohydrate intake to 5-10 % of total energy from carbohydrates, but derive at least 70 % of total energy from fat.

SUMMARY:
The study evaluates the timeline of changes of body composition, physical and psychological performance, and biochemical markers of metabolism and inflammation responses to low energy ketogenic diet for loosing weight in obese individuals. The participants will be monitored and guided by the interdisciplinary obesity team for 12 weeks.

DETAILED DESCRIPTION:
Ketogenic diets have been shown to be an effective tool to fight obesity with reported good adherence due to their ability to suppress the drive to eat. They are also gaining popularity in public, despite some concerns regarding the quality and timeline of changes of body composition and the effects on health parameters of whole organism.

For effective weight loss, energy deficit is required. Very low energy (600 - 800 kcal) ketogenic diets have been extensively studied.

The proposed study combines low energy (800 - 1500 kcal) and ketogenic diet intervention. The aim of the study is a comprehensive determination of quality of body mass loss, metabolic states changes, physical and psychological performance changes, and inflammatory and hormones profile changes during and post a 12-week low energy ketogenic diet intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2
* asymptomatic for any disease except obesity

Exclusion Criteria:

* presence of cardiovascular, endocrine, acute or chronic inflammatory diseases;
* taking medications for lipid metabolism, or psychiatric disorders;
* adherence to a prescribed diet;
* unstable weight in the past 3 months;
* BMI < 30 kg/m2;
* unwilling or unable to eat the foods prescribed in the study;
* vigorous physical activity;
* pregnancy or lactation.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-18 (Actual); Primary Completion 2017-06-17 (Actual); Study Completion 2018-06-24 (Actual)

PRIMARY OUTCOMES:
Change in body composition | Change from baseline over 12 weeks with intermediate time points at 1, 2, 4 and 8 weeks.
  Body mass, fat free body mass and fat mass will be measured (all in kilograms) with bioelectrical impedance analysis (BIA) Tanita BC 418MA.
Change in beta-hydroxybutirate | Change from baseline over 12 weeks with intermediate time points at 1, 2, 4 and 8 weeks.
  Overnight fasted serum beta-hydroxybutirate will be determined (in mmol/l).
Change in resting energy rate | Change from baseline to 12 weeks.
  Resting energy rate will be determined with indirect calorimetry.
Change in physical fitness | Change from baseline to 12 weeks.
  Physical fitness will be determined using 2 km walking test according to the UKK Walk Test Programme.
Change in cognitive functions | Change from baseline to 12 weeks.
  Will be assessed by validated psychological test (Wechsler Adult Intelligence Scale - Forth Edition (WAIS-IV).
Change in psychological factors | Change from baseline to 12 weeks.
  Will be assessed by validated psychological test (Dutch Eating Behavior Questionnaire (DEBQ).

SECONDARY OUTCOMES:
Change in body weight following intervention | Change from 12 weeks to 12 months.
  Maintenance of body mass at the end of intervention will be evaluated over the 12 months following intervention (in kilogrames).
Adherence to ketogenic diet | At 12 months.
  Adherence to ketogenic diet will be assessed by 3-day food record.

CONTACTS AND LOCATIONS:
Overall Officials: Zala Jenko Pražnikar, PhD, Principal Investigator — University of Primorska, Faculty of Health Sciences
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Noakes TD, Windt J. Evidence that supports the prescription of low-carbohydrate high-fat diets: a narrative review. Br J Sports Med. 2017 Jan;51(2):133-139. doi: 10.1136/bjsports-2016-096491. PMID 28053201
- [Background] Yang MU, Van Itallie TB. Composition of weight lost during short-term weight reduction. Metabolic responses of obese subjects to starvation and low-calorie ketogenic and nonketogenic diets. J Clin Invest. 1976 Sep;58(3):722-30. doi: 10.1172/JCI108519. PMID 956398
- [Background] Urbain P, Strom L, Morawski L, Wehrle A, Deibert P, Bertz H. Impact of a 6-week non-energy-restricted ketogenic diet on physical fitness, body composition and biochemical parameters in healthy adults. Nutr Metab (Lond). 2017 Feb 20;14:17. doi: 10.1186/s12986-017-0175-5. eCollection 2017. PMID 28239404
- [Background] Paoli A, Bianco A, Damiani E, Bosco G. Ketogenic diet in neuromuscular and neurodegenerative diseases. Biomed Res Int. 2014;2014:474296. doi: 10.1155/2014/474296. Epub 2014 Jul 3. PMID 25101284